CLINICAL TRIAL: NCT04264858
Title: An Exploratory Clinical Study on the Treatment of Acute Severe 2019-nCoV Pneumonia With Immunoglobulin From Cured 2019-nCoV Pneumonia Patients
Brief Title: Treatment of Acute Severe 2019-nCoV Pneumonia With Immunoglobulin From Cured Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiang Cheng, Head of department of cardiology, Wuhan Union Hospital, China, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WuhanUH-2019 nCoV-Ig
Record Dates: First submitted 2020-02-08; First posted 2020-02-11 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: 2019-nCoV; Immunoglobulin of Cured Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Immunoglobulin of cured patients
  Interventions: Drug: Immunoglobulin of cured patients
- Control group (Placebo Comparator): γ-Globulin
  Interventions: Drug: γ-Globulin

INTERVENTIONS:
Drug: Immunoglobulin of cured patients — 0.2g/kg, ivdrip, once a day, for 3 days
  Arms: Treatment group
Drug: γ-Globulin — 0.2g/kg, ivdrip, once a day, for 3 days
  Arms: Control group

SUMMARY:
The new coronavirus pneumonia is an acute infectious pneumonia. The pathogen is a previously unknown new coronavirus, namely 2019 new coronavirus (2019 novel coronavirus, 2019 nCoV). However, there is no specific anti-viral drug. It has been found that the specific antibodies against virus antigen are produced after these patients were cured, which could block the infection of 2019 nCoV on the host cells. At present, immunoadsorption is the most direct, rapid and effective method to separate immunoglobulin from the cured patients. Therefore, the study aims to prepare the immunoglobulin from 2019-ncov pneumonia cured patients, evaluate the efficacy and safety of the immunoglobulin in 2019-ncov pneumonia cured patients on the treatment of acute severe 2019-ncov pneumonia, and provide a new strategy for the treatment of 2019-ncov pneumonia.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteers who have understood and signed the informed consent;
2. Age ≥18 years, gender unlimited;
3. Patients diagnosed with acute severe 2019-nCoV pneumonia:

   1. Laboratory (RT-PCR) confirmed infection with 2019-nCoV.
   2. Lung involvement confirmed with pulmonary CT scan.
   3. At least one of the following conditions should be met: respiratory distress, RR ≥ 30 times/min; oxygen saturation ≤ 93% in resting state; PaO2/FiO2 ≤ 300mmHg; respiratory failure and mechanical ventilation are required; shock occurs; ICU monitoring and treatment is required in combination with other organ failure.

Exclusion Criteria:

1. Viral pneumonia with other viruses besides 2019-nCoV.
2. Patients are not suitable for immunoglobulin therapy.
3. Participation in other studies.
4. Other circumstances in which the investigator determined that the patient is not suitable for the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-03-17 (Estimated); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Time to Clinical Improvement (TTCI) | up to 28 days
  TTCI is defined as the time (in days) from initiation of study treatment (active or placebo) until a decline of two categories from admission status on a six-category ordinal scale of clinical status which ranges from 1 (discharged) to 6 (death).
  Six-category ordinal scale: 6. Death; 5. ICU, requiring ECMO and/or IMV; 4. ICU/hospitalization, requiring NIV/ HFNC therapy; 3. Hospitalization, requiring supplemental oxygen (but not NIV/ HFNC); 2. Hospitalization, not requiring supplemental oxygen; 1. Hospital discharge.
  Abbreviation: IMV, invasive mechanical ventilation; NIV, non-invasive mechanical ventilation; HFNC, High-flow nasal cannula.

SECONDARY OUTCOMES:
Clinical status assessed by the ordinal scale | up to 28 days
  on days 7, 14, 21, and 28
The differences in oxygen intake methods | up to 28 days
  1. No need for supplemental oxygenation; 2. nasal cathete oxygen inhalation；3. Mask oxygen inhalation；4. Noninvasive ventilator oxygen supply；5. Invasive ventilator oxygen supply.
Duration (days) of supplemental oxygenation | up to 28 days
Duration (days) of mechanical ventilation | up to 28 days
The mean PaO2/FiO2 | up to 28 days
The lesions of the pulmonary segment numbers involved in pulmonary CT [ every 7 days] | up to 28 days
  The detection frequency could be increased according to clinician's decision
Time to 2019-nCoV RT-PCR negativity in respiratory tract specimens [every 3 days] | up to 28 days
Dynamic changes of 2019-nCoV antibody titer in blood | up to 28 days
  The antibody titer is detected on days 3 and 28
Length of hospital stay (days) | up to 28 days
All cause mortality | up to 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China